CLINICAL TRIAL: NCT03578263
Title: Carbetocin Versus Oxytocin and Ergometrine for Prevention of Postpartum Hemorrhage Following a Cesarean Section in Women With Multiple Gestation
Brief Title: Carbetocin Versus Oxytocin and Ergometrine for the Prevention of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/204/2/18
Record Dates: First submitted 2018-05-14; First posted 2018-07-06 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; post-partum hemorrhage; multiple pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin; Ergonovine

STUDY DESIGN:
Intervention Model Description: The current study was a single-blinded randomized controlled trial conducted at a tertiary University Hospital Women included in the study were divided into 2 groups: Group (A): included 100 patients who received carbetocin 100 µg diluted in 10 ml normal saline and administered slowly (over 30-60 seconds) intravenously by anesthetist after birth of the baby. Group (B): included 100 patients who received a combination of intraoperative oxytocin 5 I.U which was diluted in 10 ml normal saline and administered slowly over (30-60 seconds) intravenously by anesthetist and intramuscular ergometrine 0.2 mg.
Who Masked: Participant
Masking Description: the participants blinded the arms of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbetocin arm (Experimental): carbetocin 100 µg diluted in 10 ml normal saline and administered slowly (over 30-60 seconds) intravenously by anesthetist after the birth of the baby
  Interventions: Drug: Carbetocin
- oxytocin and ergometrine arm (Active Comparator): oxytocin 5 I.U which was diluted in 10 ml normal saline and administered slowly over (30-60 seconds) intravenously by anesthetist plus intramuscular ergometrine 0.2 mg after the birth of the baby
  Interventions: Drug: oxytocin; Drug: ergometrine

INTERVENTIONS:
Drug: Carbetocin — Group (A): included 100 patients who received carbetocin 100 µg diluted in 10 ml normal saline and administered slowly (over 30-60 seconds) intravenously by anesthetist after the birth of the baby.
  Other Names: Pabal
  Arms: carbetocin arm
Drug: oxytocin — Group (B): included 100 patients who received a combination of intraoperative oxytocin 5 I.U which was diluted in 10 ml normal saline and administered slowly over (30-60 seconds) intravenously by anesthetist and
  Other Names: Active Comparator
  Arms: oxytocin and ergometrine arm
Drug: ergometrine — intramuscular ergometrine 0.2 mg.
  Other Names: Active Comparator
  Arms: oxytocin and ergometrine arm

SUMMARY:
The cesarean section is a bloody operation, about 750 to 1000 ml are lost at most operations and over 1000 ml of blood have lost to bring them into the definition of a postpartum hemorrhage (PPH). In developing countries, PPH is the main cause of maternal deaths. Uterine atony is the most common cause of immediate heavy PPH.Multiple pregnancy ones of a common factor for uterine atony. The administration of oxytocic's after the delivery of the neonate reduces the likelihood of PPH and 5 IU oxytocin by slow intravenous injection is currently recommended for all cesarean sections. However, the use of additional oxytocic medication is common, to arrest bleeding, or prophylactically if there are risk factors for PPH . Carbetocin is a synthetic analog of human oxytocin with structural modifications that increase its half-life, thereby prolonging its pharmacological effects. Carbetocin has been approved in 23 countries for prevention of uterine atony and excessive bleeding following cesarean delivery in spinal or epidural anesthesia. Oxytocin is a peptide of nine amino acids (Nona peptide). The structure of oxytocin is very similar to that of arginine vasopressin, whose sequence differs from oxytocin by 2 amino acids. The best-known mechanism for oxytocin to exert its stimulatory effect on myometrial contractility is by increasing the intracellular concentration of calcium. Owing to its short plasma half-life (mean 3 min), a continuous intravenous infusion is required to maintain the uterus in a contracted state. The usual dose is 20 IU in 500 ml of crystalloid solution, with the dosage rate adjusted according to response. Ergometrine is a selective and moderately potent tryptaminergic receptor antagonist in various smooth muscles, being only a partially agonistic or antagonistic at tryptaminergic receptors in the central nervous system. In blood vessels, the alkaloid is only weakly antagonistic of dopaminergic receptors and partially agonistic of α-adrenergic receptors. oxytocin (19%). Blood loss>500 ml was only observed in women who received oxytocin. The aim of the investigator's study was to compare the effect of carbetocin vs. oxytocin and ergometrine for prevention of PPH during cesarean section in women with multiple pregnancies.

DETAILED DESCRIPTION:
Women included in the study were divided into 2 groups: Group (A): included patients who received carbetocin 100 µg diluted in 10 ml normal saline and administered slowly (over 30-60 seconds) intravenously by anesthetist after the birth of the baby. Group (B): included patients who received a combination of intraoperative oxytocin 5 I.U which was diluted in 10 ml normal saline and administered slowly over (30-60 seconds) intravenously by anesthetist and intramuscular ergometrine 0.2 mg. The slow administration has been shown to reduce the potentially harmful hemodynamic effects of oxytocin (and presumably carbetocin). Also, intramuscular injection of ergometrine did the same. All women were subjected to full history taking, general and obstetric examination and investigations in the form of preoperative routine labs and obstetric ultrasound, and postoperative serum hemoglobin %.

ELIGIBILITY:
Inclusion Criteria:

* women with a multiple term pregnancy undergoing elective cesarean section

Exclusion Criteria:

* single gestation
* placenta praevia and placental abruption
* undergoing cesarean section with general anesthesia
* women undergoing cesarean section at less than 37 weeks of gestation
* with a severe medical disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 220 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
estimation of intraoperative blood loss (ml). | intraoperative
  Intraoperative blood loss was measured suction bottle and the difference in weight (in grams) between the dry and the soaked operation sheets and towels (1 gram = 1 ml.). Post-operative blood loss was measured through intraperitoneal suction drain which measured every 12 hours and on removing the drain. After that, the total blood loss was calculated by the addition of intraoperative and postoperative blood loss.and vaginal bleeding

SECONDARY OUTCOMES:
need for blood transfusion | 24 hours postoperative
  need for blood transfusion
Hemoglobin concentration | ist 24 hours postoperative]
  pre and postoperative hemoglobin estimation

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt